CLINICAL TRIAL: NCT06259682
Title: A Mixed-method Pilot Investigation of Paradoxical Intention for Insomnia. Assessing Acceptability, Feasibility and Preliminary Effectiveness.
Brief Title: A Mixed-method Pilot Investigation of Paradoxical Intention for Insomnia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-06594-01
Record Dates: First submitted 2024-01-18; First posted 2024-02-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Insomnia; Comorbidities and Coexisting Conditions
Keywords: Insomnia disorder; mechanisms; mixed-methods; paradoxical intention; sleep performance anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Uncontrolled pilot study using mixed methods investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): Only one arm, all participants are given the treatment
  Interventions: Behavioral: Paradoxical Intention

INTERVENTIONS:
Behavioral: Paradoxical Intention — Paradoxical intention (PI). PI is described as instructing patients with sleep onset insomnia to try to remain awake for as long as possible rather than to focus on trying to fall asleep

SUMMARY:
The investigators aim to test the preliminary efficacy as well as the acceptability and feasibility of paradoxical intention, which is a psychotherapeutic technique, for improving insomnia symptoms in adults. Previous research has tested this technique for insomnia and found overall positive results. However, during the last decades very few studies have examined paradoxical intention. Therefore the investigators wish to conduct a pilot study examining the effects in a modern context.

DETAILED DESCRIPTION:
In the 1970s, Ascher and Efran developed paradoxical intention (PI), instructing sleep onset insomnia patients to stay awake instead of trying to sleep. The American Academy of Sleep Medicine confirmed PI's effectiveness. However, between 2006-2018, PI use in clinical practice declined.

The study will investigate PI's acceptability, mechanisms, and predictors for effectiveness. It involves a pilot trial with 40 insomnia patients in Sweden, recruited through advertisements and screened through web questionnaires, phone interviews, and sleep diaries. Criteria are based on insomnia research standards and Diagnostic and Statistical Manual Fifth Edition (DSM-5), including insomnia with common comorbidities.

Participants will undergo baseline assessments, then receive four weekly online PI modules, including educational texts, behavioral experiments, and homework. Weekly therapist meetings via phone or video will support and troubleshoot issues.

Post-treatment, 10-15 participants will be randomly selected for qualitative interviews to evaluate their experiences with PI, focusing on sleep patterns, text volume, therapist support, and homework's impact on sleep quality and treatment adherence. Interviews will be audio-recorded and analyzed thematically.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing three screening phases: a web-based questionnaire, a telephone interview with a structured assessment, and a 7-day sleep diary completion.
* Screening resulting in diagnosis of insomnia, including co-morbid insomnia.
* Participant should fulfill the following DSM-5 criteria. (1)Difficulty in sleep Initiation, maintenance, or early morning awakening. (2)Frequency and duration of at least three nights per week and has been present for at least three months.(3) Problems persist despite candidates having had adequate opportunity and circumstances for sleep. (4) The sleep disturbance causes significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning.
* Age above 18 and Swedish resident and language proficient.

Exclusion Criteria:

* Severe depressive episode with suicidal intentions or actions
* Current or past diagnosis of psychotic or bipolar disorders
* Current substance use disorder
* Recent changes in psychopharmacotherapy (within the last three months) or use of "as-needed" hypnotic medications during the trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline (Week 0). Weekly assessments every week for four weeks, with a final assessment following the fourth and final module (total duration of 4 weeks). Follow-up assessment at 12 weeks post-treatment completion
  Measure of severity of insomnia

SECONDARY OUTCOMES:
Sleep diary | Baseline (Week 0). One assessment at week 2 of treatment program following second module and one at week 4 following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Idiographic sleep diary
Work and Social Adjustment Scale (WSAS) | Baseline (Week 0). One assessment at week 4 of treatment program following the completion of the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of functional impairment
Depression Anxiety Stress Scales (DASS) | Baseline (Week 0). One assessment at week 2 of treatment program following second module and one at week 4 following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of depressive anxiety symptoms
Brunnsviken Brief Quality of Life Scale (BBQ | Baseline (Week 0). One assessment at week 4 of treatment program following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of quality of life.

OTHER OUTCOMES:
Sleep Anxiety Scale (SAS) | Baseline (Week 0). One assessment at week 2 of treatment program following second module and one at week 4 following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of anticipatory anxiety before bedtime
Glasgow Sleep Effort Scale (GSES) | Baseline (Week 0). One assessment at week 2 of treatment program following second module and one at week 4 following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of sleep effort exerted.
Metacognitions Questionnaire - Insomnia (MCQ-I) | Baseline (Week 0). One assessment at week 2 of treatment program following second module and one at week 4 following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of metacognitions around sleep.
Sleep Problem Acceptance Questionnaire (SPAQ) | Baseline (Week 0). One assessment at week 2 of treatment program following second module and one at week 4 following the fourth and final module. Follow-up assessment at 12 weeks post-treatment completion
  Measure of acceptance of sleep issues
Client Satisfaction Questionnaire (CSQ) | One assessment at week 4 of treatment program following the fourth and final module.
  Measure of satisfaction of treatment.
Credibility/Expectancy Questionnaire (CEQ) | Once at week 1 of treatment (immediately following module 1)
  Credibility and expectancy measure for participant to answer
Negative effects Questionnaire (NEQ) | Once at week 4 of treatment (immediately following fourth and final module)
  Measure of clients experience of negative effects during therapy

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Karolinska Institutet, Stockholm
  - Karolinska Institute, Stockholm
  - Örebro University, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salim O, Jansson-Frojmark M, Sandlund C, Norell A. Paradoxical intention as a treatment for insomnia disorder: study protocol for a mixed-methods pilot trial. BMJ Open. 2024 Oct 10;14(10):e086676. doi: 10.1136/bmjopen-2024-086676. PMID 39389596